CLINICAL TRIAL: NCT01132313
Title: Safety, Antiviral Effect and Pharmacokinetics of BI 207127 in Combination With BI 201335 and With or Without Ribavirin for 4, 16, 24, 28 or 40 Weeks in Patients With Chronic HCV Genotype 1 Infection (Randomized Phase Ib/II)
Brief Title: Safety, Antiviral Effect and PK of BI 207127 + BI 201335 +/- RBV for 4 up to 40 Weeks in Patients With Chronic HCV Genotype 1 Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1241.21; 2009-018197-66 (EudraCT Number: EudraCT)
Record Dates: First submitted 2010-05-03; First posted 2010-05-28 (Estimated); Results first posted 2016-02-01 (Estimated); Last update posted 2016-02-01 (Estimated); Status verified 2015-12

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — deleobuvir; faldaprevir; Ribavirin

ARMS (12):
- 2 (Experimental): 4 weeks of high dose TID BI 207127 and QD BI 201335 in combination with RBV, Part 1
  Interventions: Drug: Ribavirin; Drug: BI 201335; Drug: BI 207127
- 1 (Experimental): 4 weeks of low dose three times per day (TID) BI 207127 and once daily (QD) BI 201335 in combination with RBV, Part 1
  Interventions: Drug: BI 207127; Drug: BI 201335; Drug: Ribavirin
- 3 (Experimental): 16 weeks of TID BI 207127 and QD BI 201335 in combination with RBV, Part 2
  Interventions: Drug: BI 207127; Drug: BI 201335; Drug: Ribavirin
- 4 (Experimental): 28 weeks of TID BI 207127 and QD BI 201335 in combination with RBV, Part 2
  Interventions: Drug: BI 207127; Drug: Ribavirin; Drug: BI 201335
- 5 (Experimental): 40 weeks of TID BI 207127 and QD BI 201335 in combination with RBV, Part 2
  Interventions: Drug: BI 201335; Drug: BI 207127; Drug: Ribavirin
- 6 (Experimental): 28 weeks of BID BI 207127 and QD BI 201335 in combination with RBV, Part 2
  Interventions: Drug: Ribavirin; Drug: BI 201335; Drug: BI 207217
- 7 (Experimental): 28 weeks of TID BI 207127 and QD BI 201335 without RBV, Part 2
  Interventions: Drug: BI 207127; Drug: BI 201335
- 8 (Experimental): 16 weeks of BID BI 207127 and QD BI 201335 in combination with RBV, Part 3
  Interventions: Drug: BI 207127; Drug: Ribavirin; Drug: BI 201335
- 9 (Experimental): 24 weeks of BID BI 207127 and QD BI 201335 in combination with RBV, Part 3
  Interventions: Drug: BI 207127; Drug: BI 201335; Drug: Ribavirin
- 10 (Experimental): 24 weeks of TID BI 207127 and QD BI 201335 in combination with RBV, Part 3
  Interventions: Drug: BI 201335; Drug: BI 207127; Drug: Ribavirin
- 11 (Experimental): 16 weeks of BID BI 207127 and QD BI 201335 in combination with RBV, Part 4
  Interventions: Drug: Ribavirin; Drug: BI 207127; Drug: BI 201335
- 12 (Experimental): 24 weeks of BID BI 207127 and QD BI 201335 in combination with RBV, Part 4
  Interventions: Drug: Ribavirin; Drug: BI 201335; Drug: BI 207127

INTERVENTIONS:
Drug: BI 207127 — 28 weeks, high dose, TID
  Arms: 4
Drug: BI 201335 — 40 weeks, QD
  Arms: 5
Drug: BI 207127 — 4 weeks, low dose TID
  Arms: 1
Drug: BI 201335 — 24 weeks, QD
  Arms: 1
Drug: Ribavirin — 16 weeks, according to label
  Arms: 11
Drug: Ribavirin — 28 weeks, according to label
  Arms: 4
Drug: Ribavirin — 28 weeks, according to label
  Arms: 6
Drug: BI 207127 — 40 weeks, high dose, TID
  Arms: 5
Drug: BI 207127 — 24 weeks, very high dose, BID
  Arms: 9
Drug: BI 207127 — 16 weeks, standard dose, BID
  Arms: 11
Drug: BI 201335 — 24 weeks, QD
  Arms: 10
Drug: Ribavirin — 48 weeks, according to label
  Arms: 2
Drug: Ribavirin — 40 weeks, according to label
  Arms: 5
Drug: BI 207127 — 16 weeks, high dose, TID
  Arms: 3
Drug: BI 207127 — 28 weeks, high dose, TID
  Arms: 7
Drug: BI 201335 — 28 weeks, QD
  Arms: 6
Drug: BI 201335 — 16 weeks, QD
  Arms: 11
Drug: Ribavirin — 24 weeks, according to label
  Arms: 12
Drug: BI 201335 — 24 weeks, QD
  Arms: 12
Drug: BI 201335 — 28 weeks, QD
  Arms: 7
Drug: BI 207127 — 24 weeks, standard dose, BID
  Arms: 12
Drug: BI 201335 — 24 weeks, QD
  Arms: 9
Drug: BI 201335 — 16 weeks, QD
  Arms: 3
Drug: BI 207127 — 16 weeks, high dose, BID
  Arms: 8
Drug: BI 201335 — 24 weeks, QD
  Arms: 2
Drug: Ribavirin — 16 weeks, according to label
  Arms: 3
Drug: Ribavirin — 16 weeks, according to label
  Arms: 8
Drug: BI 207217 — 28 weeks, high dose BID
  Arms: 6
Drug: BI 201335 — 16 weeks, QD
  Arms: 8
Drug: BI 207127 — 24 weeks, high dose, TID
  Arms: 10
Drug: Ribavirin — 48 weeks, according to label
  Arms: 1
Drug: BI 207127 — 4 weeks, high dose, TID
  Arms: 2
Drug: BI 201335 — 28 weeks, QD
  Arms: 4
Drug: Ribavirin — 24 weeks, according to label
  Arms: 9
Drug: Ribavirin — 24 weeks, according to label
  Arms: 10

SUMMARY:
The substances BI 201335 and BI 207127 are being developed for the treatment of chronic hepatitis C virus infection. BI 201335 and BI 207127 work by preventing the virus from replicating.

The currently available medications pegylated interferon alfa and ribavirin for hepatitis C ca have considerable adverse events in patients and in many cases are not sufficiently effective. This is particularly the case in treatment of patients infected with genotype 1 of HCV.

A combination therapy of these new substances without pegylated interferon alfa may be associated with fewer adverse events that currently available (pegylated interferon-alfa-based) medication and may also provide a treatment option to the large number of patients with contraindications or intolerance to pegylated interferon alfa.

This clinical trial (1241.21) currently consists of 3 distinct studies: Part 1, Part 2 and Part 3.

Part 1 (SOUND-C1) is a 2 armed study as described in experimental arms 1 and 2 below (actual enrollment: 56 patients; randomized and treated: 32) Part 2 (SOUND-C2) is a 5 armed study as described in experimental arms 3 to 7 below (actual enrollment: 465; randomized and treated: 362) Part 3 (SOUND-C3) includes 3 arms as described in experimental arms 8 to 10 below (83 patients randomized and treated)

ELIGIBILITY:
Inclusion criteria:

* Chronic hepatitis C virus (HCV) infection of genotype (GT) 1
* Parts 1-3:Treatment naive to Interferon -alfa (IFN), Pegylated interferon -alfa (PegIFN), ribavirin (RBV), and any direct acting antiviral agent for chronic hepatitis C
* Part 4: Treatment experienced with confirmed prior virological failure to an approved dose of PegIFN/RBV (null-response)
* HCV RNA >=10,000 IU/mL at screening
* Liver biopsy within two years or fibroscan within six months prior to baseline
* Liver biopsy within two years or fibroscan within 6 months prior to screening
* Age 18-75 years

Exclusion criteria:

* Hepatitis C virus (HCV) infection of mixed genotype
* Evidence of liver disease due to causes other than chronic HCV infection
* Positive ELISA for human immunodeficiency virus (HIV)
* Hepatitis B virus (HBV) infection
* Decompensated liver disease or history of decompensated liver disease
* Active or suspected malignancy within the last 5 years
* Ongoing or historical photosensitivity or recurrent rash
* History of alcohol or drug abuse (except cannabis) within the past 12 months
* Body mass index (BMI)I <18 or > 35 kg/m2
* Usage of any investigational drugs within 30 days prior to enrolment, or 5 half-lives, whichever is longer; o the planned usage of an investigational drug during the course of the current study
* Known hypersensitivity to any ingredient of the study drugs
* A condition that is defined as one which in the opinion of the investigator may interfere with the patient's capability for participation in the trial or may influence the results of the trial
* Alpha fetoprotein >100ng/mL at screening; if >20ng/mL and <=100ng/mL, patients can be included if there is no evidence of liver cancer in an appropriate imaging study within 6 months prior to randomisation
* Total bilirubin > 2 mg/dL with ratio of direct/indirect > 1
* AST or ALT >5xULN
* INR prolonged to >1.7xULN
* Requirement for chronic systemic corticosteroids
* Received concomitant systemic antiviral, hematopoietic growth factor, or immunomodulatory treatment within 30 days prior to enrolment or 5 half-lives, whichever is longer
* Received silymarin or glycyrrhizin or Sho-saiko-to within 30 days prior to enrolment
* Contraindications pertaining to PegIFN or RBV

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 488 (Actual)
Dates: Start 2010-05; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (53):
- United States (12):
  - 1241.21.0003 Boehringer Ingelheim Investigational Site, La Jolla, California
  - 1241.21.0006 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1241.21.0004 Boehringer Ingelheim Investigational Site, San Francisco, California
  - 1241.21.0011 Boehringer Ingelheim Investigational Site, Palm Harbor, Florida
  - 1241.21.0013 Boehringer Ingelheim Investigational Site, Valparaiso, Indiana
  - 1241.21.0008 Boehringer Ingelheim Investigational Site, Springfield, Massachusetts
  - 1241.21.0019 Boehringer Ingelheim Investigational Site, Fayetteville, North Carolina
  - 1241.21.0012 Boehringer Ingelheim Investigational Site, Arlington, Texas
  - 1241.21.0005 Boehringer Ingelheim Investigational Site, Austin, Texas
  - 1241.21.0007 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1241.21.0010 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1241.21.0017 Boehringer Ingelheim Investigational Site, Seattle, Washington
- Australia (2):
  - 1241.21.61002 Boehringer Ingelheim Investigational Site, Heidelberg, Victoria
  - 1241.21.61001 Boehringer Ingelheim Investigational Site, Melbourne, Victoria
- Austria (3):
  - 1241.21.43003 Boehringer Ingelheim Investigational Site, Linz
  - 1241.21.43001 Boehringer Ingelheim Investigational Site, Vienna
  - 1241.21.43002 Boehringer Ingelheim Investigational Site, Vienna
- France (8):
  - 1241.21.33005 Boehringer Ingelheim Investigational Site, Clichy
  - 1241.21.33007 Boehringer Ingelheim Investigational Site, Grenoble Cédex 9
  - 1241.21.33003 Boehringer Ingelheim Investigational Site, Lyon
  - 1241.21.33001 Boehringer Ingelheim Investigational Site, Marseille
  - 1241.21.33002 Boehringer Ingelheim Investigational Site, Montpellier
  - 1241.21.33004 Boehringer Ingelheim Investigational Site, Paris
  - 1241.21.33008 Boehringer Ingelheim Investigational Site, Paris
  - 1241.21.33006 Boehringer Ingelheim Investigational Site, Vandœuvre-lès-Nancy
- Germany (9):
  - 1241.21.49002 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.21.49003 Boehringer Ingelheim Investigational Site, Berlin
  - 1241.21.49007 Boehringer Ingelheim Investigational Site, Düsseldorf
  - 1241.21.49005 Boehringer Ingelheim Investigational Site, Esslingen am Neckar
  - 1241.21.49001 Boehringer Ingelheim Investigational Site, Frankfurt am Main
  - 1241.21.49006 Boehringer Ingelheim Investigational Site, Hamburg
  - 1241.21.49009 Boehringer Ingelheim Investigational Site, Hanover
  - 1241.21.49004 Boehringer Ingelheim Investigational Site, Leipzig
  - 1241.21.49008 Boehringer Ingelheim Investigational Site, Mainz
- 1241.21.64001 Boehringer Ingelheim Investigational Site, Auckland NZ, New Zealand
- Portugal (5):
  - 1241.21.35103 Boehringer Ingelheim Investigational Site, Aveiro
  - 1241.21.35104 Boehringer Ingelheim Investigational Site, Coimbra
  - 1241.21.35101 Boehringer Ingelheim Investigational Site, Lisbon
  - 1241.21.35105 Boehringer Ingelheim Investigational Site, Lisbon
  - 1241.21.35102 Boehringer Ingelheim Investigational Site, Porto
- Romania (3):
  - 1241.21.40001 Boehringer Ingelheim Investigational Site, Bucharest
  - 1241.21.40002 Boehringer Ingelheim Investigational Site, Bucharest
  - 1241.21.40003 Boehringer Ingelheim Investigational Site, Bucharest
- Spain (6):
  - 1241.21.34002 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.21.34005 Boehringer Ingelheim Investigational Site, Barcelona
  - 1241.21.34003 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.21.34004 Boehringer Ingelheim Investigational Site, Madrid
  - 1241.21.34001 Boehringer Ingelheim Investigational Site, Majadahonda-Madrid
  - 1241.21.34006 Boehringer Ingelheim Investigational Site, Valencia
- Switzerland (4):
  - 1241.21.41003 Boehringer Ingelheim Investigational Site, Basel
  - 1241.21.41006 Boehringer Ingelheim Investigational Site, Bern
  - 1241.21.41001 Boehringer Ingelheim Investigational Site, Sankt Gallen
  - 1241.21.41002 Boehringer Ingelheim Investigational Site, Zurich

REFERENCES:
- [Derived] Zeuzem S, Mantry P, Soriano V, Buynak RJ, Dufour JF, Pockros PJ, Wright D, Angus P, Buti M, Stern JO, Kadus W, Vinisko R, Bocher W, Mensa FJ. Short article: Faldaprevir, deleobuvir and ribavirin in IL28B non-CC patients with HCV genotype-1a infection included in the SOUND-C3 phase 2b study. Eur J Gastroenterol Hepatol. 2016 Aug;28(8):923-6. doi: 10.1097/MEG.0000000000000649. PMID 27140229
- [Derived] Asselah T, Zeuzem S, Soriano V, Bronowicki JP, Lohse AW, Mullhaupt B, Schuchmann M, Bourliere M, Buti M, Roberts SK, Gane EJ, Stern JO, Voss F, Baum P, Gallivan JP, Bocher WO, Mensa FJ. ITPA Genotypes Predict Anemia but Do Not Affect Virological Response with Interferon-Free Faldaprevir, Deleobuvir, and Ribavirin for HCV Infection. PLoS One. 2015 Dec 9;10(12):e0144004. doi: 10.1371/journal.pone.0144004. eCollection 2015. PMID 26650626
- [Derived] Zeuzem S, Soriano V, Asselah T, Gane EJ, Bronowicki JP, Angus P, Lohse AW, Stickel F, Mullhaupt B, Roberts S, Schuchmann M, Manns M, Bourliere M, Buti M, Stern JO, Gallivan JP, Voss F, Sabo JP, Bocher W, Mensa FJ; SOUND-C2 Study Group. Efficacy and safety of faldaprevir, deleobuvir, and ribavirin in treatment-naive patients with chronic hepatitis C virus infection and advanced liver fibrosis or cirrhosis. Antimicrob Agents Chemother. 2015 Feb;59(2):1282-91. doi: 10.1128/AAC.04383-14. Epub 2014 Dec 15. PMID 25512403
- [Derived] Zeuzem S, Soriano V, Asselah T, Bronowicki JP, Lohse AW, Mullhaupt B, Schuchmann M, Bourliere M, Buti M, Roberts SK, Gane EJ, Stern JO, Vinisko R, Kukolj G, Gallivan JP, Bocher WO, Mensa FJ. Faldaprevir and deleobuvir for HCV genotype 1 infection. N Engl J Med. 2013 Aug 15;369(7):630-9. doi: 10.1056/NEJMoa1213557. PMID 23944300
- [Derived] Zeuzem S, Asselah T, Angus P, Zarski JP, Larrey D, Mullhaupt B, Gane E, Schuchmann M, Lohse AW, Pol S, Bronowicki JP, Roberts S, Arasteh K, Zoulim F, Heim M, Stern JO, Nehmiz G, Kukolj G, Bocher WO, Mensa FJ. Faldaprevir (BI 201335), deleobuvir (BI 207127) and ribavirin oral therapy for treatment-naive HCV genotype 1: SOUND-C1 final results. Antivir Ther. 2013;18(8):1015-9. doi: 10.3851/IMP2567. Epub 2013 Apr 4. PMID 23558093

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: This trial was conducted in 4 parts, each consisting of randomised, open-label treatments.
Groups:
- Part 1: 400mg DBV and 120mg FDV - 4w: Part 1: 4 weeks of 400mg Deleobuvir tablet TID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. From week 5 to week 24, patients received treatment with FDV 120mg QD in combination with standard of care (SOC) PegIFN/RBV (triple therapy period)
- Part 1: 600mg DBV and 120mg FDV - 4w: Part 1: 4 weeks of 600mg Deleobuvir (DBV, BI 207127) tablet three times per day (TID) and 120mg Faldaprevir (FDV, BI 201335) soft gelatin capsule once daily (QD) in combination with Ribavirin (RBV) tablet. From week 5 to week 24, patients received treatment with FDV 120mg QD in combination with SOC PegIFN/RBV (triple therapy period)
- Part 2: 600mg DBV and 120mg FDV - 16w: Part 2: 16 weeks of 600mg Deleobuvir tablet TID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 2: 600mg DBV TID and 120mg FDV - 28w: Part 2: 28 weeks of 600mg Deleobuvir tablet TID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 2: 600mg DBV and 120mg FDV - 40w: Part 2: 40 weeks of 600mg Deleobuvir tablet TID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 2: 600mg DBV BID and 120mg FDV - 28w: Part 2: 28 weeks of 600mg Deleobuvir tablet twice a day (BID) and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 2: 600mg DBV and 120mg FDV, no RBV - 28w: Part 2: 28 weeks of 600mg Deleobuvir tablet TID and 120mg Faldaprevir soft gelatin capsule QD, without RBV. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 3: 600mg DBV and 120mg FDV - 16w: Part 3: 16 weeks of 600mg Deleobuvir tablet BID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 3: 800mg DBV and 120mg FDV - 24w: Part 3: 24 weeks of 800mg Deleobuvir tablet BID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 3: 600mg DBV and 120mg FDV - 24w: Part 3: 24 weeks of 600mg Deleobuvir tablet TID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet. Patients who discontinued their assigned treatment early due to lack of antiviral activity could receive additional treatment with PegIFN/RBV for up to 24 weeks.
- Part 4: 600 mg DBV and 120mg FDV - 16w: Part 4: 16 weeks of 600mg Deleobuvir tablet BID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet.
- Part 4: 600 mg DBV and 120mg FDV - 24w: Part 4: 24 weeks of 600mg Deleobuvir tablet BID and 120mg Faldaprevir soft gelatin capsule QD in combination with RBV tablet.
Period: Overall Study
Arm/Group | Part 1: 400mg DBV and 120mg FDV - 4w | Part 1: 600mg DBV and 120mg FDV - 4w | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w | Part 3: 600mg DBV and 120mg FDV - 16w | Part 3: 800mg DBV and 120mg FDV - 24w | Part 3: 600mg DBV and 120mg FDV - 24w | Part 4: 600 mg DBV and 120mg FDV - 16w | Part 4: 600 mg DBV and 120mg FDV - 24w
Started | 17 | 17 | 81 | 80 | 79 | 79 | 49 | 32 | 26 | 25 | 1 | 2
Completed | 14 | 17 | 61 | 48 | 34 | 54 | 19 | 24 | 5 | 5 | 0 | 2
Not Completed | 3 | 0 | 20 | 32 | 45 | 25 | 30 | 8 | 21 | 20 | 1 | 0
Not completed — Lack of Efficacy | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 3 | 14 | 16 | 0 | 0
Not completed — Not treated | 2 | 0 | 0 | 0 | 2 | 1 | 3 | 0 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 0 | 0 | 4 | 10 | 19 | 6 | 5 | 3 | 7 | 2 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 0 | 3 | 3 | 6 | 0 | 1 | 0 | 0 | 2 | 0 | 0
Not completed — Lack of antiviral response | 0 | 0 | 12 | 18 | 18 | 18 | 21 | 0 | 0 | 0 | 1 | 0
Not completed — Other reason not defined above | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Treated set which included all patients who were dispensed study medication and were documented to have taken at least one dose of investigational treatment regardless of randomisation.
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: 400mg DBV and 120mg FDV - 4w | Part 1: 600mg DBV and 120mg FDV - 4w | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w | Part 3: 600mg DBV and 120mg FDV - 16w | Part 3: 800mg DBV and 120mg FDV - 24w | Part 3: 600mg DBV and 120mg FDV - 24w | Part 4: 600 mg DBV and 120mg FDV - 16w | Part 4: 600 mg DBV and 120mg FDV - 24w | Total
Number analyzed (Participants) | 15 | 17 | 81 | 80 | 77 | 78 | 46 | 32 | 26 | 25 | 1 | 2 | 480
Age, Continuous [Mean (Standard Deviation); unit: Years] | 50.8 (10.0) | 50.8 (11.5) | 48.6 (11.3) | 47.3 (11.2) | 48.9 (10.7) | 47.9 (11.1) | 45.3 (13.0) | 48.9 (11.8) | 47.2 (13.4) | 46.5 (12.5) | 59.0 (NA) — Not calculable due to only one patient in treatment group | 52.5 (4.9) | 48.1 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 7 | 36 | 39 | 41 | 37 | 22 | 20 | 11 | 11 | 1 | 2 | 234
  Male | 8 | 10 | 45 | 41 | 36 | 41 | 24 | 12 | 15 | 14 | 0 | 0 | 246

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Rapid Virological Response (RVR)
Description: Part 1: Rapid virological response (RVR), defined as Hepatitis C Virus Ribonucleic acid (HCV RNA) <25IU/mL at Week 4 of treatment
Time Frame: 4 weeks
Population: FAS which included all randomised patients who were dispensed study medication and were documented to have taken at least one dose of study medication.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 1: 400mg DBV and 120mg FDV - 4w | Part 1: 600mg DBV and 120mg FDV - 4w
Number analyzed (Participants) | 15 | 17
Percentage of participants | 73.3 [47.6 to 89.0] | 100.0 [84.7 to 100.0]

2. Primary Outcome: Part 2: Sustained Virological Response (SVR)
Description: Part 2: Sustained virological response (SVR), defined as HCV RNA <25 IU/mL and undetectable at 12 weeks after end of treatment
Time Frame: From drug administration until 12 weeks after end of treatment, up to 52 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w
Number analyzed (Participants) | 81 | 80 | 77 | 78 | 46
Percentage of participants | 59.3 | 58.8 | 51.9 | 69.2 | 39.1

3. Primary Outcome: Part 3 and 4: Sustained Virological Response (SVR)
Description: Part 3 and 4: Sustained virological response (SVR) defined as HCV RNA <25IU/mL and undetectable at 12 weeks after end of treatment
Time Frame: From drug administration until 12 weeks after end of treatment, up to 36 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 3: 600mg DBV and 120mg FDV - 16w | Part 3: 800mg DBV and 120mg FDV - 24w | Part 3: 600mg DBV and 120mg FDV - 24w | Part 4: 600 mg DBV and 120mg FDV - 16w | Part 4: 600 mg DBV and 120mg FDV - 24w
Number analyzed (Participants) | 32 | 26 | 25 | 1 | 2
Percentage of participants | 65.6 [46.8 to 81.4] | 19.2 [6.6 to 39.4] | 12.0 [2.5 to 31.2] | NA [NA to NA] — The study was stopped before data were collected from the participants in Part 4 | NA [NA to NA] — The study was stopped before data were collected from the participants in Part 4

4. Secondary Outcome: Part 1: Time to Virological Response
Description: Part 1: Time to virological response, defined as the timepoint of the first measurement of plasma HCV RNA level <25 IU/mL. The percentage of participants who achieved virological response within each time period are displayed for this outcome measure.
Time Frame: From drug administration until end of drug administration, up to 4 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: 400mg DBV and 120mg FDV - 4w | Part 1: 600mg DBV and 120mg FDV - 4w
Number analyzed (Participants) | 15 | 17
Percentage of participants
  <= 2 weeks | 6.7 | 11.8
  <= 4 weeks | 20.0 | 47.1
  <= 8 weeks | 53.3 | 41.2
  <= 12 weeks | 0.0 | 0.0
  <= 16 weeks | 6.7 | 0.0
  <= 28 weeks | 0.0 | 0.0
  <= 32 weeks | 6.7 | 0.0
  <= 40 weeks | 0.0 | 0.0
  > 40 weeks | 0.0 | 0.0
  Never | 6.7 | 0.0

5. Secondary Outcome: Part 2: Time to Virological Response
Description: Part 2: Time to virological response, defined as the timepoint of the first measurement of plasma HCV RNA level <25 IU/mL. The percentage of participants who achieved virological response within each time period are displayed for this outcome measure.
Time Frame: From drug administration until end of drug administration, up to 40 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w
Number analyzed (Participants) | 81 | 80 | 77 | 78 | 46
Percentage of participants
  Day 0 (N=81, 80, 77, 78, 46) | 0.0 | 0.0 | 0.0 | 0.0 | 0.0
  Day 8(N=75, 72, 72, 75, 44) | 3.8 | 7.7 | 1.4 | 2.6 | 2.2
  Day 15 (N=62, 61, 63, 60, 33) | 19.4 | 20.7 | 9.9 | 22.1 | 19.3
  Day 29 (N=29, 32, 27, 32, 21) | 61.5 | 55.5 | 59.4 | 57.7 | 48.6
  Day 43 (N=16, 12, 13, 18, 12) | 78.8 | 83.3 | 80.5 | 76.2 | 70.7
  Day 57 (N=9, 8, 9, 11, 9) | 88.1 | 88.9 | 85.1 | 85.5 | 78.0
  Day 85 (N=9, 7, 8, 11, 9) | 88.1 | 90.3 | 86.8 | 85.5 | 78.0
  Day 113 (N=9, 7, 8, 11, 8) | 88.1 | 90.3 | 86.8 | 85.5 | 80.4
  Day 141 (N=9, 7, 8, 11, 8) | 88.1 | 90.3 | 86.8 | 85.5 | 80.4
  Day 169 (N=9, 7, 8, 11, 8) | 88.1 | 90.3 | 86.8 | 85.5 | 80.4
  Day 197 (N=9, 7, 8, 11, 8) | 88.1 | 90.3 | 86.8 | 85.5 | 80.4

6. Secondary Outcome: Part 1 and 2: Plasma HCV RNA Level Not Detectable at Week 4
Description: Part 1 and 2: Plasma Hepatitis C Virus Ribonucleic acid (HCV RNA) level not detectable at Week 4
Time Frame: 4 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Part 1: 400mg DBV and 120mg FDV - 4w | Part 1: 600mg DBV and 120mg FDV - 4w | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w
Number analyzed (Participants) | 15 | 17 | 81 | 80 | 77 | 78 | 46
Percentage of participants | 20.0 | 70.6 | 65.4 | 60.0 | 63.6 | 56.4 | 50.0

7. Secondary Outcome: Part 2: Sustained Virological Response at 4 and 24 Weeks After End of Treatment
Description: Part 2: Sustained virological response at 4 and 24 weeks after end of treatment
Time Frame: 4 weeks and 24 weeks after the end of treatment, up to 64 weeks
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w
Number analyzed (Participants) | 81 | 80 | 77 | 78 | 46
Percentage of participants
  SVR4 | 60.5 | 62.5 | 54.5 | 69.2 | 43.5
  SVR24 | 58.0 | 58.8 | 49.4 | 69.2 | 39.1

8. Secondary Outcome: Part 3 and 4: Plasma HCV RNA Level <25 IU/mL at Week 4 and 12 of Treatment
Description: Part 3 and 4: Plasma Hepatitis C Virus Ribonucleic acid (HCV RNA) level <25 IU/mL at week 4 and 12 of treatment
Time Frame: Week 4 and 12
Population: FAS
Measure: Number; unit: Percentage of participants
Arm/Group | Part 3: 600mg DBV and 120mg FDV - 16w | Part 3: 800mg DBV and 120mg FDV - 24w | Part 3: 600mg DBV and 120mg FDV - 24w | Part 4: 600 mg DBV and 120mg FDV - 16w | Part 4: 600 mg DBV and 120mg FDV - 24w
Number analyzed (Participants) | 32 | 26 | 25 | 1 | 2
Percentage of participants | 75.0 | 26.9 | 32.0 | NA — The study was stopped before data were collected from the participants in Part 4 | NA — The study was stopped before data were collected from the participants in Part 4

9. Secondary Outcome: Part 3 and 4: Sustained Virological Response (SVR) at 4 Weeks After End of Treatment
Description: Part 3 and 4: Sustained virological response (SVR) at 4 weeks after end of treatment
Time Frame: up to 28 weeks
Population: FAS
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Part 3: 600mg DBV and 120mg FDV - 16w | Part 3: 800mg DBV and 120mg FDV - 24w | Part 3: 600mg DBV and 120mg FDV - 24w | Part 4: 600 mg DBV and 120mg FDV - 16w | Part 4: 600 mg DBV and 120mg FDV - 24w
Number analyzed (Participants) | 32 | 26 | 25 | 1 | 2
Percentage of participants | 75.0 [56.6 to 88.5] | 19.2 [6.6 to 39.4] | 12.0 [2.5 to 31.2] | NA [NA to NA] — The study was stopped before data were collected from the participants in Part 4 | NA [NA to NA] — The study was stopped before data were collected from the participants in Part 4

ADVERSE EVENTS:
Time Frame: From first drug administration until 30 days after last drug administration for parts 1, 2 and 4 and until 28 days after last drug administration for part 3, up to 361 days
Arm/Group | Part 1: 400mg DBV and 120mg FDV - 4w | Part 1: 600mg DBV and 120mg FDV - 4w | Part 2: 600mg DBV and 120mg FDV - 16w | Part 2: 600mg DBV TID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV - 40w | Part 2: 600mg DBV BID and 120mg FDV - 28w | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w | Part 3: 600mg DBV and 120mg FDV - 16w | Part 3: 800mg DBV and 120mg FDV - 24w | Part 3: 600mg DBV and 120mg FDV - 24w | Part 4: 600 mg DBV and 120mg FDV - 16w | Part 4: 600 mg DBV and 120mg FDV - 24w
Serious Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 3/81 | 8/80 | 6/77 | 8/78 | 3/46 | 1/32 | 3/26 | 2/25 | 0/1 | 0/2
Other Adverse Events (participants affected / at risk) | 0/15 | 0/17 | 76/81 | 71/80 | 74/77 | 73/78 | 43/46 | 30/32 | 26/26 | 25/25 | 1/1 | 2/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 400mg DBV and 120mg FDV - 4w (N=15) | Part 1: 600mg DBV and 120mg FDV - 4w (N=17) | Part 2: 600mg DBV and 120mg FDV - 16w (N=81) | Part 2: 600mg DBV TID and 120mg FDV - 28w (N=80) | Part 2: 600mg DBV and 120mg FDV - 40w (N=77) | Part 2: 600mg DBV BID and 120mg FDV - 28w (N=78) | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w (N=46) | Part 3: 600mg DBV and 120mg FDV - 16w (N=32) | Part 3: 800mg DBV and 120mg FDV - 24w (N=26) | Part 3: 600mg DBV and 120mg FDV - 24w (N=25) | Part 4: 600 mg DBV and 120mg FDV - 16w (N=1) | Part 4: 600 mg DBV and 120mg FDV - 24w (N=2)
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Accident at work (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Angina unstable (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0
B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Blood potassium decreased (Investigations) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Brain injury (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Bundle branch block left (Cardiac disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cardiopulmonary failure (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Cellulitis pharyngeal (Infections and infestations) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Coronary artery disease (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Coronary artery stenosis (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Electrocardiogram QT prolonged (Investigations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Erythema nodosum (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Febrile neutropenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Gun shot wound (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Limb traumatic amputation (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Myocardial infarction (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Prerenal failure (Renal and urinary disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0
Psychotic disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Purpura (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Retinal tear (Eye disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Toxic skin eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1 | 0 | 1 | 0 | 0 | 0 | 0 | 0
Ventricular fibrillation (Cardiac disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 1 | 0 | 0 | 0 | 0 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Part 1: 400mg DBV and 120mg FDV - 4w (N=15) | Part 1: 600mg DBV and 120mg FDV - 4w (N=17) | Part 2: 600mg DBV and 120mg FDV - 16w (N=81) | Part 2: 600mg DBV TID and 120mg FDV - 28w (N=80) | Part 2: 600mg DBV and 120mg FDV - 40w (N=77) | Part 2: 600mg DBV BID and 120mg FDV - 28w (N=78) | Part 2: 600mg DBV and 120mg FDV, no RBV - 28w (N=46) | Part 3: 600mg DBV and 120mg FDV - 16w (N=32) | Part 3: 800mg DBV and 120mg FDV - 24w (N=26) | Part 3: 600mg DBV and 120mg FDV - 24w (N=25) | Part 4: 600 mg DBV and 120mg FDV - 16w (N=1) | Part 4: 600 mg DBV and 120mg FDV - 24w (N=2)
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 1 | 6 | 0 | 4 | 2 | 2 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 0 | 0 | 4 | 3 | 7 | 4 | 3 | 1 | 1 | 0 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 7 | 7 | 6 | 12 | 8 | 0 | 3 | 3 | 0 | 0
Abdominal pain upper (Gastrointestinal disorders) | 0 | 0 | 6 | 15 | 12 | 2 | 2 | 3 | 5 | 2 | 0 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 7 | 2 | 7 | 4 | 1 | 2 | 0 | 0 | 0
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 1 | 9 | 10 | 7 | 0 | 8 | 3 | 2 | 1 | 0
Anxiety (Psychiatric disorders) | 0 | 0 | 3 | 4 | 7 | 4 | 0 | 2 | 2 | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 5 | 4 | 4 | 3 | 0 | 1 | 0 | 0 | 0
Asthenia (General disorders) | 0 | 0 | 24 | 28 | 25 | 21 | 7 | 7 | 4 | 1 | 0 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 3 | 3 | 1 | 6 | 0 | 1 | 1 | 1 | 0 | 0
Chest pain (General disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 0 | 1 | 0 | 1
Chills (General disorders) | 0 | 0 | 5 | 2 | 3 | 2 | 2 | 1 | 1 | 0 | 0 | 0
Constipation (Gastrointestinal disorders) | 0 | 0 | 4 | 1 | 6 | 3 | 1 | 4 | 4 | 1 | 0 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 7 | 4 | 10 | 9 | 2 | 2 | 2 | 2 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 4 | 15 | 10 | 8 | 0 | 3 | 0 | 1 | 0 | 0
Depressed mood (Psychiatric disorders) | 0 | 0 | 1 | 2 | 5 | 2 | 0 | 0 | 1 | 0 | 0 | 0
Depression (Psychiatric disorders) | 0 | 0 | 1 | 10 | 5 | 5 | 1 | 0 | 2 | 2 | 0 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 34 | 33 | 36 | 29 | 12 | 7 | 9 | 9 | 0 | 0
Disturbance in attention (Nervous system disorders) | 0 | 0 | 3 | 4 | 4 | 3 | 3 | 1 | 1 | 0 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 4 | 3 | 5 | 3 | 1 | 5 | 1 | 3 | 0 | 1
Dry eye (Eye disorders) | 0 | 0 | 0 | 0 | 3 | 1 | 0 | 2 | 0 | 0 | 0 | 0
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 4 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 12 | 12 | 11 | 18 | 7 | 3 | 2 | 2 | 0 | 0
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 4 | 5 | 2 | 2 | 0 | 2 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 0 | 0 | 6 | 5 | 8 | 14 | 4 | 6 | 4 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 8 | 10 | 4 | 0 | 0 | 1 | 0 | 0 | 1
Eczema (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 3 | 2 | 4 | 3 | 0 | 1 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1 | 4 | 1 | 0 | 0 | 1 | 0 | 0 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 1 | 1 | 3 | 0 | 0
Fatigue (General disorders) | 0 | 0 | 18 | 14 | 22 | 21 | 7 | 9 | 9 | 10 | 1 | 0
Flatulence (Gastrointestinal disorders) | 0 | 0 | 3 | 5 | 4 | 4 | 2 | 2 | 1 | 1 | 0 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 0 | 0 | 4 | 2 | 2 | 0 | 1 | 2 | 2 | 0 | 1
Headache (Nervous system disorders) | 0 | 0 | 11 | 8 | 15 | 11 | 7 | 4 | 3 | 2 | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 0 | 0 | 2 | 3 | 0 | 0 | 3 | 0 | 0 | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 2 | 0 | 0 | 1 | 3 | 0 | 0
Hypoaesthesia oral (Gastrointestinal disorders) | 0 | 0 | 0 | 1 | 0 | 0 | 1 | 1 | 0 | 2 | 0 | 0
Influenza like illness (General disorders) | 0 | 0 | 2 | 6 | 5 | 5 | 2 | 0 | 0 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 11 | 8 | 12 | 7 | 2 | 4 | 3 | 5 | 0 | 0
Irritability (General disorders) | 0 | 0 | 8 | 6 | 4 | 2 | 1 | 0 | 1 | 2 | 0 | 0
Jaundice (Hepatobiliary disorders) | 0 | 0 | 25 | 22 | 15 | 16 | 2 | 6 | 5 | 4 | 0 | 0
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 1 | 2 | 1 | 1 | 2 | 0 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 0 | 0 | 1 | 2 | 1 | 1 | 4 | 0 | 0 | 1 | 0 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 4 | 1 | 6 | 3 | 1 | 1 | 2 | 1 | 0 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 4 | 4 | 3 | 1 | 2 | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 4 | 8 | 7 | 6 | 6 | 2 | 0 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 0 | 41 | 43 | 41 | 39 | 26 | 18 | 16 | 18 | 1 | 1
Ocular icterus (Eye disorders) | 0 | 0 | 2 | 0 | 3 | 5 | 0 | 2 | 2 | 1 | 0 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 1 | 2 | 3 | 1 | 1 | 2 | 1 | 0 | 0
Pain of skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 1
Papule (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 2 | 1 | 0 | 0 | 0
Paraesthesia (Nervous system disorders) | 0 | 0 | 10 | 9 | 6 | 4 | 5 | 0 | 3 | 2 | 0 | 0
Photosensitivity reaction (Skin and subcutaneous tissue disorders) | 0 | 0 | 20 | 23 | 23 | 19 | 11 | 4 | 3 | 8 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 0 | 16 | 24 | 31 | 23 | 14 | 7 | 6 | 7 | 0 | 2
Pyrexia (General disorders) | 0 | 0 | 1 | 4 | 4 | 4 | 1 | 1 | 2 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 21 | 11 | 28 | 15 | 13 | 0 | 9 | 10 | 0 | 2
Rash papulosquamous (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 1 | 0 | 0 | 0
Sleep disorder (Psychiatric disorders) | 0 | 0 | 3 | 4 | 7 | 4 | 2 | 0 | 1 | 0 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 1 | 4 | 0 | 0 | 0
Sunburn (Injury, poisoning and procedural complications) | 0 | 0 | 6 | 4 | 9 | 6 | 8 | 1 | 2 | 4 | 0 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1 | 2 | 5 | 6 | 0 | 0 | 0 | 0 | 0 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 2 | 0 | 0 | 0 | 0
Tremor (Nervous system disorders) | 0 | 0 | 0 | 1 | 1 | 1 | 1 | 2 | 0 | 1 | 0 | 0
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 2 | 0 | 2 | 1 | 2 | 0 | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 24 | 29 | 23 | 20 | 13 | 11 | 6 | 5 | 0 | 0
Weight decreased (Investigations) | 0 | 0 | 8 | 6 | 11 | 8 | 4 | 0 | 2 | 2 | 0 | 0

LIMITATIONS AND CAVEATS:
There were only 3 patients entered in part 4 of the trial, therefore no formal analyses of efficacy data were performed.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.